CLINICAL TRIAL: NCT01060111
Title: Adequate Therapy of Topiramate in Migraine
Brief Title: An Efficacy and Tolerability Study of Topiramate in Participants With Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR011944; MIG-KOR-001
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Results first posted 2013-08-06 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Migraine
Keywords: Migraine; Topiramate; Propranolol
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Topiramate Standard (Experimental): Topiramate 25 mg will be administered once daily and the dose will be increased by 25 mg per day at an interval of 1-week up to a dose of 50 mg to 100 mg up to Week 6. A maintenance dose of 50 mg to 100 mg will be administered twice daily up to Week 10 as per Physician's discretion.
  Interventions: Drug: Topiramate Standard
- Topiramate Slow (Experimental): Topiramate 25 mg will be administered once daily and the dose will be increased by 25 mg per day at an interval of 2-weeks up to a dose of 50 mg to 100 mg up to Week 6. A maintenance dose of 50 mg to 100 mg will be administered twice daily up to Week 10 as per Physician's discretion.
  Interventions: Drug: Topiramate Slow
- Topiramate Slow and Propranolol Booster (Experimental): Topiramate 25 mg will be administered once daily and the dose will be increased by 25 mg per day at an interval of 2-weeks up to a dose of 50 mg to 100 mg up to Week 6. A maintenance dose of 50 mg to 100 mg will be administered twice daily up to Week 10 as per Physician's discretion. Propranolol 80 mg will be administered once daily, 40 mg in the morning and 40 mg in the evening up to Week 6.
  Interventions: Drug: Topiramate Slow; Drug: Propranolol booster

INTERVENTIONS:
Drug: Topiramate Standard — Topiramate 25 mg will be administered once daily and the dose will be increased by 25 mg per day at an interval of 1-week up to a dose of 50 mg to 100 mg up to Week 6. A maintenance dose of 50 mg to 100 mg will be administered twice daily up to Week 10 as per Physician's discretion.
  Arms: Topiramate Standard
Drug: Topiramate Slow — Topiramate 25 mg will be administered once daily and the dose will be increased by 25 mg per day at an interval of 2-weeks up to a dose of 50 mg to 100 mg up to Week 6. A maintenance dose of 50 mg to 100 mg will be administered twice daily up to Week 10 as per Physician's discretion.
  Arms: Topiramate Slow; Topiramate Slow and Propranolol Booster
Drug: Propranolol booster — Propranolol 80 mg will be administered once daily, 40 mg in the morning and 40 mg in the evening up to Week 6.
  Arms: Topiramate Slow and Propranolol Booster

SUMMARY:
The purpose of this study is to investigate the adequacy (reasonably good) of topiramate therapy (medicine or medical care given to a participant for a disease or condition) in prevention of migraine (type of severe headache that occurs periodically and is often associated with nausea, vomiting, and constipation or diarrhea) by comparing standard titration (slow increase in drug dosage, guided by patient's responses) therapy to slow titration therapy and slow titration therapy boosted by the concurrent use of propranolol in participants with migraine with or without aura (having to do with the ear) for more than or equal to 2 attacks per month.

DETAILED DESCRIPTION:
This is a prospective (study following participants forward in time), single-blind (Physician does not know the intervention), randomized (study drug assigned by chance) and comparative multi-center (conducted in more than 1 center) study to assess appropriate administration methods with topiramate preventive therapy in participants with migraine. The study consists of 3 periods: Screening period (4 weeks), Treatment period consisting of 2 titration periods (3 weeks each) and Maintenance period (4 weeks). During Screening period, after the diagnosis of participants' headache, symptoms and severity of migraine will be investigated through a headache diary and participants will be selected for treatment period. In the treatment period, the selected participants will be randomly assigned to either of the 3 topiramate therapy: 'topiramate standard group', 'topiramate slow group', and 'topiramate slow plus propranolol (booster) group'. In the 'topiramate standard group' - participants will receive an initial dose of topiramate 25 milligram (mg) once daily and the dose of topiramate will be increased by 25 mg per day at an interval of 1-week up to the target dose of 50 mg to 100 mg up to Week 6; and a maintenance dose of 50 mg to 100 mg will be administered twice daily up to Week 10 as per Physician's discretion. In 'topiramate slow group' - participants will start with an initial dose of 25 mg once daily and the dose will be increased by 25 mg per day at an interval of 2-weeks up to a dose of 50 mg to 100 mg up to Week 6. A maintenance dose of 50 mg to 100 mg will be administered twice daily up to Week 10 as per Physician's discretion. In 'topiramate slow plus propranolol (booster) group' - participants will follow the same dosage regimen as in the 'topiramate slow group' along with concurrent administration of booster dose of propranolol 80 mg once daily (40 mg each time in the morning and in the evening) for 6 weeks. The participants will primarily be evaluated for reduction in migraine frequency between Week 7 and 10 using a headache diary questionnaire maintained by them. Participants' quality of life will be assessed using Migraine Disability Assessment (MIDAS) score and intensity of pain in migraine will be assessed using Visual Analogue Scale (VAS). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Particpants who have signed the consent form
* Participants who have 3 to 14 episodes of migraine a month
* Participants whose duration of migraine is at least 6 months
* Participants who can read and understand the migraine disability assessment (MIDAS) questionnaire
* Female Participants who are using an appropriate contraception method or have negative pregnancy test results

Exclusion Criteria:

* Participants whose headache attacks at Baseline or during the study period are assumed to be caused by a drug withdrawal syndrome
* Participants whose migraine has appeared first at over 50 years of age
* Participants who have taken anticonvulsants (valproic acid, gabapentin), beta adrenergic blockers (propranolol) and calcium antagonists (sibelium, verapamil, diltiazem) or topiramate or propranolol within the last 8 weeks
* Participants with progressive neurological (pertaining to the nervous system) disorder
* Participants with severe renal (pertaining to the kidneys) disorder, hepatic (pertaining to the liver) failure or diabetes (disorder in which there is decreased insulin in the body or the body's insulin is not effective, resulting in high blood sugar, increased thirst and urine, and many other side effects) or with the history of renal calculus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2006-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (6):
- South Korea (6):
  - Busan
  - Daegu
  - Kwangjoo
  - Kyunggi-Do
  - Seoul
  - Uijeongbu-si

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 250 consented participants, 243 participants were assigned to study treatment.
Groups:
- Topiramate Standard: Topiramate 25 milligram (mg) was administered once daily and the dose was increased by 25 mg per day at an interval of 1-week up to a dose of 50 mg to 100 mg up to Week 6. A maintenance dose of 50 mg to 100 mg was administered twice daily up to Week 10 as per Physician's discretion.
- Topiramate Slow: Topiramate 25 mg was administered once daily and the dose was increased by 25 mg per day at an interval of 2-weeks up to a dose of 50 mg to 100 mg up to Week 6. A maintenance dose of 50 mg to 100 mg was administered twice daily up to Week 10 as per Physician's discretion.
- Topiramate Slow and Propranolol Booster: Topiramate 25 mg was administered once daily and the dose was increased by 25 mg per day at an interval of 2-weeks up to a dose of 50 mg to 100 mg up to Week 6. A maintenance dose of 50 mg to 100 mg was administered twice daily up to Week 10 as per Physician's discretion. Propranolol 80 mg was administered once daily, 40 mg in the morning and 40 mg in the evening up to Week 6.
Period: Overall Study
Arm/Group | Topiramate Standard | Topiramate Slow | Topiramate Slow and Propranolol Booster
Started | 81 | 84 | 80
Treated | 81 | 83 | 79
Completed | 54 | 61 | 45
Not Completed | 27 | 23 | 35
Not completed — Adverse Event | 9 | 5 | 18
Not completed — Lack of Efficacy | 2 | 1 | 0
Not completed — Inappropriate participant | 5 | 4 | 5
Not completed — Participants' evasion for hospital visit | 0 | 3 | 2
Not completed — Participants' non-cooperation | 8 | 6 | 6
Not completed — Adverse event and insufficient effect | 0 | 1 | 0
Not completed — Participants' non-cooperation | 1 | 0 | 0
Not completed — Other | 2 | 3 | 4

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were measured for Intent-to-treat (ITT) population which was defined as participants who took topiramate at least once and had migraine improvement data at the Week 6.
Groups:
- Topiramate Standard: Topiramate 25 mg was administered once daily and the dose was increased by 25 mg per day at an interval of 1-week up to a dose of 50 mg to 100 mg up to Week 6. A maintenance dose of 50 mg to 100 mg was administered twice daily up to Week 10 as per Physician's discretion.
- Total: Total of all reporting groups
Arm/Group | Topiramate Standard | Topiramate Slow | Topiramate Slow and Propranolol Booster | Total
Number analyzed (Participants) | 81 | 83 | 78 | 242
Age, Customized [Number; unit: Participants] — Age, Customized was measured for ITT population which was defined as participants who took topiramate at least once and had migraine improvement data at the Week 6. Here 'N=239' (80, 82, and 78 for topiramate standard, topiramate slow, topiramate slow and propranolol booster groups respectively) signifies the participants who were evaluated for this Baseline characteristic.
  Participants
    Age 20 and over but younger than age 30 | 16 | 23 | 22 | 61
    Age 30 and over but younger than age 40 | 24 | 27 | 30 | 81
    Age 40 and over but younger than age 50 | 22 | 19 | 16 | 57
    Age 50 and over but younger than age 60 | 11 | 11 | 7 | 29
    Age 60 and over | 7 | 2 | 2 | 11
Sex: Female, Male [Count of Participants; unit: Participants] — Gender was measured for ITT population which was defined as participants who took topiramate at least once and had migraine improvement data at the Week 6.
  Participants
    Female | 72 | 76 | 63 | 211
    Male | 9 | 7 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Percentage Decrease in Migraine Episodes
Description: Decrease in percentage of migraine frequency (episodes) was measured from baseline using a headache diary which is a typical scale measuring neuropsychiatric symptoms in a migraine participant. Migraine will be diagnosed in accordance with the guidelines of the International Headache Society (IHS).
Time Frame: Maintenance period (Weeks 7 to 10)
Population: The intent-to-treat (ITT) population included all the participants who took topiramate at least once and had migraine improvement data at the Week 6. Here 'N' signifies participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage decrease in migraine episodes
Arm/Group | Topiramate Standard | Topiramate Slow | Topiramate Slow and Propranolol Booster
Number analyzed (Participants) | 51 | 57 | 43
Percentage decrease in migraine episodes | 48 (69) | 57 (48) | 46 (69)
Statistical Analysis 1: Comparison: Topiramate Standard vs Topiramate Slow vs Topiramate Slow and Propranolol Booster; Test type: Superiority or Other; p = 0.6207, ANOVA; Analysis of Variance (ANOVA) for treatment groups (Topiramate standard, Topiramate slow, Topiramate slow and Propranolol booster) was used
Statistical Analysis 2: Comparison: Topiramate Standard vs Topiramate Slow and Propranolol Booster; Test type: Non-Inferiority or Equivalence — Non-inferioirity was to be concluded if the ratio of percentage decrease in migraine episodes was greater than 0.7. Power of calculation was 0.9, significance level was 0.025; p = 0.5, t-test, 1 sided; Ratio of percentage decrease = 0.950, 95% CI 2-sided [0.519 to 1.737]

2. Secondary Outcome: Change From Baseline in Migraine Frequency at Week 6
Description: The migraine frequency at Week 6 was evaluated through a headache diary completed by a participant and the reduction rate of migraine frequency compared to the Baseline period was measured. Change values were calculated as Baseline value minus value at Week 6.
Time Frame: Baseline and Week 6
Population: The ITT population included all the participants who took topiramate at least once and had migraine improvement data at the Week 6. Here 'n' signifies participants evaluable for this outcome measure at given time point.
Measure: Mean (Standard Deviation); unit: Migraine episodes/Week
Groups:
- Topiramate Standard: Topiramate Capsule 25 mg administered once daily till week 1. From Week 2 dose was increased by 25 mg every Week till a dose of 50 mg to 100 mg up to Week 6 and a dose of 50 mg to 100 mg twice daily up to Week 10 as per Physician's discretion.
- Topiramate Slow: Topiramate Capsule 25 mg administered once daily till week 1. From Week 2 dose was increased by 25 mg every 2 Weeks till a dose of 50 mg to 100 mg up to Week 6 and a dose of 50 mg to 100 mg twice daily up to Week 10 as per Physician's discretion.
- Topiramate Slow and Propranolol Booster: Topiramate Capsule 25 mg administered once daily till week 1. From Week 2 dose was increased by 25 mg every 2 Weeks till a dose of 50 mg to 100 mg up to Week 6 and a dose of 50 mg to 100 mg twice daily up to Week 10 as per Physician's discretion. Propranolol 80 mg administered once daily, 40 mg in the morning and 40 mg in the evening up to Week 6.
Arm/Group | Topiramate Standard | Topiramate Slow | Topiramate Slow and Propranolol Booster
Number analyzed (Participants) | 81 | 83 | 78
Migraine episodes/Week
  Baseline | 1.48 (0.76) | 1.58 (0.80) | 1.59 (0.87)
  Change at Week 6 (n=51, 57, 43) | 0.89 (1.04) | 0.89 (0.88) | 0.74 (1.31)
Statistical Analysis 1: Comparison: Topiramate Standard vs Topiramate Slow vs Topiramate Slow and Propranolol Booster; Test type: Superiority or Other; p = 0.7247, ANOVA; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Migraine Disability Assessment (MIDAS) Score at Week 6
Description: MIDAS scoring ranges from 0 to 63. The scores are divided into ranges of disability with higher scores indicating increased disability as follows: 0-5 (Grade I - Minimal or infrequent disability); 6-10 (Grade II - Mild or infrequent disability); 11-20 (Grade III - Moderate disability); and 21+ (Grade IV - Severe disability). Change values were calculated as Baseline value minus value at Week 6.
Time Frame: Baseline and Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Topiramate Standard | Topiramate Slow | Topiramate Slow and Propranolol Booster
Number analyzed (Participants) | 81 | 83 | 78
Units on a scale
  Baseline | 1.32 (1.26) | 1.29 (1.14) | 1.42 (1.77)
  Change at Week 6 (n=54, 61, 44) | 0.99 (1.18) | 0.99 (1.08) | 0.95 (2.00)
Statistical Analysis 1: Comparison: Topiramate Standard vs Topiramate Slow vs Topiramate Slow and Propranolol Booster; Test type: Superiority or Other; p = 0.9872, ANOVA; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score at Week 6
Description: VAS was used to measure the intensity of migraine. The assessment scale ranges from 0 to 10. One end of the line drawn on the questionnaire is marked with 0 point indicating "no headache" and the other end with 10 points indicating "unimaginably strong headache." It means that the higher the score, the severe the pain is. Change values were calculated as Baseline value minus value at Week 6.
Time Frame: Baseline and Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Topiramate Standard | Topiramate Slow | Topiramate Slow and Propranolol Booster
Number analyzed (Participants) | 81 | 82 | 76
Units on a Scale
  Baseline | 5.83 (1.55) | 5.68 (1.68) | 5.51 (1.78)
  Change at Week 6 (n= 53, 59, 42) | 1.83 (2.54) | 2.45 (2.84) | 2.31 (2.32)
Statistical Analysis 1: Comparison: Topiramate Standard vs Topiramate Slow vs Topiramate Slow and Propranolol Booster; Test type: Superiority or Other; p = 0.4326, ANOVA — Analysis of Variance (ANOVA) for treatment groups (Topiramate standard, Topiramate slow, Topiramate slow and Propranolol booster) was used

ADVERSE EVENTS:
Time Frame: Baseline up to Week 10
Description: Participants evaluable for safety were 81, 83, and 79 for topiramate standard, topiramate slow, topiramate slow and propranolol booster groups respectively.
Arm/Group | Topiramate Standard | Topiramate Slow | Topiramate Slow and Propranolol Booster
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/83 | 0/79
Other Adverse Events (participants affected / at risk) | 62/81 | 62/83 | 54/79
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Topiramate Standard (N=81) | Topiramate Slow (N=83) | Topiramate Slow and Propranolol Booster (N=79)
Paresthesia (Nervous system disorders) | 42 | 48 | 36
Dizziness (Nervous system disorders) | 5 | 9 | 14
Paraesthesia (Nervous system disorders) | 6 | 5 | 3
Somnolence (Nervous system disorders) | 3 | 3 | 7
Gastrointestinal disorder (Gastrointestinal disorders) | 6 | 5 | 11
Nausea (Gastrointestinal disorders) | 1 | 2 | 5
Weight decreased (Investigations) | 14 | 7 | 9
Fatigue (General disorders) | 3 | 5 | 4
Feeling abnormal (General disorders) | 2 | 5 | 0
Anorexia (Metabolism and nutrition disorders) | 5 | 3 | 8
Psychomotor retardation (Psychiatric disorders) | 1 | 3 | 8
Depression (Psychiatric disorders) | 5 | 0 | 0
Headache (Nervous system disorders) | 7 | 5 | 3
Dyspepsia (Gastrointestinal disorders) | 4 | 0 | 1
Insomnia (Psychiatric disorders) | 4 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI cannot provide any trial related information to external parties' without mutual agreement with the Sponsor. This is valid even after the contract is cancelled.